CLINICAL TRIAL: NCT05027906
Title: A Phase 1b, Multicenter, Open Label Study to Evaluate the Safety, Pharmacokinetics and Efficacy of AT 1501 in Patients Undergoing Kidney Transplant
Brief Title: Safety, Pharmacokinetics, and Efficacy of AT 1501 in Patients Undergoing Kidney Transplant
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eledon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-1501-K102; 2021-003830-36 (EudraCT Number)
Record Dates: First submitted 2021-08-19; First posted 2021-08-30 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Prevention of Rejection in Kidney Transplant
Keywords: Kidney Transplant; Renal Allograft Rejection; Prophylaxis; AT-1501; CD40L inhibitor; Humanized blocking antibody to CD40L; Monoclonal Antibody; Renal; Transplant; ESRD; tegoprubart
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Phase 1b, open label, single-arm study
Masking Description: None ( Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AT-1501 Single Arm (Experimental): AT-1501 monoclonal antibody targeting CD40L given as an IV infusion
  Interventions: Drug: AT-1501

INTERVENTIONS:
Drug: AT-1501 — Investigative Arm

SUMMARY:
This study will evaluate the safety, PK, and efficacy of AT 1501 in patients undergoing kidney transplantation.

DETAILED DESCRIPTION:
This study will evaluate the safety, PK, and efficacy of AT 1501 in patients undergoing kidney transplantation. Up to 48 de novo kidney transplant recipients will receive AT-1501 in combination with rATG induction with corticosteroids (CS), and mycophenolate as maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Recipient of their first kidney transplant from a living or deceased donor
3. Agree to comply with contraception requirements during and for at least 90 days after the last administration of study drug

Exclusion Criteria:

1. Induction therapy, other than study assigned rATG, planned as part of initial immunosuppressive regimen
2. Currently treated with any systemic immunosuppressive regimen, including immunologic biologic therapies, with the exception of 5 mg prednisone or equivalent daily;
3. Previous treatment with AT 1501 or any other anti CD40LG therapy
4. The patient has previously received a bone marrow transplant or any other solid organ transplant, including a kidney, or will be undergoing a multi organ or dual kidney transplant
5. Will receive a kidney with an anticipated cold ischemia time of > 30 hours;
6. Will receive a kidney from a donor that meets any of the following criteria:

   * Donation after Cardiac Death (DCD) criteria; or
   * Extended Criteria Donor (ECD) criteria, defined as:
   * Is blood group (ABO) incompatible; or
   * Age ≥ 60 years; or Age 50-59 years with any 2 of the following criteria:
   * Death due to cerebrovascular accident
   * History of hypertension
   * Terminal creatinine ≥ 133 μmol/L (1.5 mg/dL)
7. Human leukocyte antigen identical (two haplotype match or zero HLA mismatch) donor
8. Medical conditions that require chronic use of systemic steroids at a dose higher than 5 mg prednisone or equivalent per day
9. History of a TE event, known hypercoagulable state, or condition requiring long term anticoagulation:
10. Positive T- or B-cell crossmatch that is due to HLA antibodies or presence of a DSA at Screening

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Safety Incidences | Through study completion, an average up to 20 months
  Incidence of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), and Adverse Events of Special Interest (AESIs)
Pharmacokinetic- PK profile | Day 1 and at steady state Month 3
  PK profile of the first dose of AT 1501 and at steady state Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (Ct), calculated using noncompartmental analysis (AUC0-t)
Pharmacokinetic- Area under the plasma concentration | Day 1 and at steady state Month 3
  Area under the plasma concentration versus time curve from time 0 extrapolated to infinity, calculated using noncompartmental analysis (AUC0-inf)
Pharmacokinetic- Cmax | Day 1 and at steady state Month 3
  Maximum observed plasma concentration (Cmax)
Pharmacokinetic- Tmax | Day 1 and at steady state Month 3
  Time to reach maximum observed plasma concentration (Tmax)
Pharmacokinetic- Ke | Day 1 and at steady state Month 3
  Terminal elimination rate constant (Ke)
Pharmacokinetic- (t1/2) | Day 1 and at steady state Month 3
  Terminal phase half-life (t1/2)
Pharmacokinetic- CL | Day 1 and at steady state Month 3
  Clearance (CL)
Pharmacokinetic- (Vdss) | Day 1 and at steady state Month 3
  Volume of distribution at steady state (Vdss)

CONTACTS AND LOCATIONS:
Locations (9):
- University of Cincinnati, Cincinnati, Ohio, United States
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Fundação Oswaldo Ramos - Hospital do Rim, São Paulo, Brazil
- Canada (3):
  - Providence Health Care - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - McGill University Health Care Centre, Montreal, Quebec
- United Kingdom (2):
  - Liverpool University Hospitals NHS Foundation Trust - Royal Liverpool University Hospital, Liverpool
  - Oxford University Hospitals NHS Foundation Trust - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No